CLINICAL TRIAL: NCT02462252
Title: A Phase IIA, Open-label Study Designed to Evaluate Efficacy and Safety of BL-8040 Followed by Anti-Thymocyte Globulin (hATG), Cyclosporine and Methylprednisolone in Adult Subjects With Aplastic Anemia (AA) or Hypoplastic Myelodysplastic Syndrome (MDS)
Brief Title: Phase IIA Open Label Study to Evaluate Efficacy and Safety of BL-8040 Followed by (hATG), Cyclosporine and Methyprednisolone in Adult Subjects With Aplastic Anemia or Hypoplastic Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioLineRx, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-8040.06
Record Dates: First submitted 2015-05-25; First posted 2015-06-04 (Estimated); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Aplastic Anemia; Hypoplastic Myelodysplastic Syndrome
MeSH Terms: conditions — Anemia, Aplastic | interventions — 4-fluorobenzoyl-TN-14003; Antilymphocyte Serum; Methylprednisolone; Methylprednisolone Hemisuccinate; Methylprednisolone Acetate; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BL-8040 plus hATG, methylprednisolone, cyclosporine (Experimental): BL-8040 0.75mg/kg will be administered Subcutaneously (SC ) on Days 1-10, then on first 5 days of months 2-6.
  Standard therapy: hATG: Days 11-14: 40mg/kg/day IV over 6-8 hours, in all AA subjects, or in MDS subjects less than 55 years old. 35mg/kg/day IV over 6-8 hours in MDS subjects 55 years and older.
  Standard therapy: methylprednisolone: Days 11-14: 40mg/kg/day IV over 6-8 hours, in all AA subjects, or in MDS subjects less than 55 years old. 35mg/kg/day IV over 6-8 hours in MDS subjects 55 years and older.
  Standard therapy: cyclosporine: 5mg/kg/day orally, given in 2 divided doses, starting on day 11 and continuing through Month 6 Day 30 (end of treatment)
  Interventions: Drug: BL-8040; Drug: horse anti-thymocyte globulin (hATG); Drug: Methylprednisolone; Drug: Cyclosporine

INTERVENTIONS:
Drug: BL-8040 — Subjects will receive subcutaneous (SC) injections of BL-8040 monotherapy on days 1-10 of the study. Beginning on Month 2 day 1, (M2/D1), and continuing monthly through Month 6, BL-8040 will be administered daily as part of the maintenance period for the first 5 days of each month.
Drug: horse anti-thymocyte globulin (hATG) — From Day 11 through Day 14 of first month, subjects will receive hATG infusion over 6-8 hours each day.
  Other Names: ATGAM
Drug: Methylprednisolone — From Day 11-14 of first month, subjects receive infusion of methylprednisolone 30 minutes prior to hATG infusion. Treatment with methylprednisolone will continue for 30 days. (After day 14, subjects may receive oral prednisone dose equivalent to IV methylprednisolone dose. The oral dose will be tapered off over 30 days.
  Other Names: Medrol, Solu-Medrol, Depo-Medrol
Drug: Cyclosporine — From Day 11 through end of treatment (Month 6 Day 30), subjects will receive oral dose of cyclosporine.
  Other Names: Sandimmune, Cyclosporine A

SUMMARY:
An open label single arm study to assess efficacy and safety of BL-8040 on top of standard immunotherapy regimen of hATG, cyclosporine and steroids in patients with Hypoplastic MDS and AA over the course of a six month (180 day) treatment period.

DETAILED DESCRIPTION:
This will be an open-label, single arm, phase IIa study in subjects with AA or Hypoplastic MDS.

Eligible subjects will receive subcutaneous (SC) injections of BL-8040 monotherapy over 10 days. From Day 11 through Day 14, subjects will receive hATG, Methylprednisolone and Cyclosporine. From Day 15 until Day 30 (of the first month), subjects will continue treatment only with Methylprednisolone and Cyclosporine. Cyclosporine will continue daily through Month 6/Day 30 (M6/D30) (end of study treatment). Beginning on M2/D1, BL-8040 will be administered daily as part of the maintenance period for the first 5 days of each month through M6. All BL-8040 injection courses will be given at the site, as either an inpatient or outpatient per the treating physician's decision.

The primary objective of the study is to determine the efficacy of the treatment with BL-8040 on top of the standard immunotherapy regimen of: hATG, cyclosporine, and steroids in patients with Hypoplastic MDS and AA. Safety and efficacy will be assessed at defined time-points throughout the study. Duration of response and overall survival will be assessed as a part of the long term FU. A maximum of 25 patients will be enrolled in the study. Subjects will be equally distributed between the disease populations.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women aged 18 and older
2. Patient must have the ability to understand the requirements of the study and provide informed consent.
3. Patients with the diagnosis of severe AA, who are not currently candidates for an allogeneic stem cell transplant, fulfilling the following criteria:

   1. BM cellularity < 30% and
   2. Peripheral blood (PB) showing at least two of the following criteria:

   Absolute neutrophil count (ANC) < 0.5 k/µL Platelet count < 30 k/µL Absolute reticulocyte count < 60,000/µL
4. Patients with recurrent/relapsed AA will be eligible for the trial as long as they were not previously refractory to hATG-based therapy and the relapse occurred > 3 months after response.
5. Patients with Hypoplastic MDS defined as MDS with marrow cellularity of:

   * < 30% for patients < 60 years,
   * < 20% for patients ≥ 60yrs.
6. Patients must have been off of cytotoxic, immunosuppressive (except steroids), or targeted therapy, including standard and investigational treatments for AA, for at least 1 week or 5 half-lives whichever comes later, prior to entering this study, and have recovered from the toxic effects of that therapy to Grade 1 or less.
7. Adequate organ function as defined below:

   • Liver function:

   a. Total bilirubin < 2.0 mg/dL (34 µmol/L) b. AST and/or ALT <3 x ULN
   * Kidney function: creatinine < 2.5 x ULN.
8. ECOG performance status of ≤ 2.
9. Women of childbearing potential and all men must agree to use an approved form of contraception (e.g. oral, transdermal patch, implanted contraceptives, intrauterine device, diaphragm, condom, abstinence or surgical sterility) prior to study entry and for the duration of study participation through 30 days after the last dose of the last treatment drug. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
10. Subject is able and willing to comply with the requirements of the protocol.
11. Subject or a legal guardian is able to voluntarily provide written informed consent.

Exclusion Criteria:

* 1. Known allergy or hypersensitivity to any of the test compounds, materials or contraindication to test product.

  2. Patients who have had any major surgical procedure within 14 days of Day 1. BM biopsy is not considered a major surgical procedure.

  3. Pregnant women are excluded from this study because the agents used in this study have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with these agents, breastfeeding should be discontinued if the mother is being treated on this trial.

  4. Seropositive for HIV antibodies (HIV1 and HIV2), Hepatitis C antibody (Hep C Ab) or a Hepatitis B carrier (positive for Hepatitis B surface antigen [HBsAg]).

  5. Life expectancy of ≤ 2 months. 6. Subjects with a clinically significant or unstable medical or surgical condition or any other condition that cannot be well-controlled by the allowed medications permitted in the study protocol that would preclude safe and complete study participation, as determined by medical history, physical examinations, ECG, laboratory tests or chest X-ray. Such conditions may include:

  • Unstable cardiovascular conditions at Baseline including but not limited to:
  * Symptomatic ischemia, or
  * Uncontrolled clinically significant conduction abnormalities (e.g., ventricular tachycardia on antiarrhythmic agents are excluded; 1st degree atrioventricular (AV) block or asymptomatic left anterior fascicular block/right bundle branch block (LAFB/RBBB) will not be excluded); or
  * Congestive heart failure (CHF) NYHA Class ≥ 3, or
  * Myocardial infarction (MI) within 3 months. • Presence of active, uncontrolled infection. • Known central nervous system illness (e.g., Alzheimer's disease).

    * A gastrointestinal disorder that may affect the absorption of study medication.
    * Use of alcohol or drug use that may interfere with the patient's ability to participate in the study.
    * Unstable psychiatric disorder that would render the patient unable to comply with study requirements.
    * Any malignancies in the 3 years prior to Baseline, excluding basal cell carcinoma, in situ malignancy, low-risk prostate cancer, cervical cancer after curative therapy.
    * A co-morbid condition that, in the Investigator's opinion, renders the subject at high risk for treatment complications.

      7. Unable to comply with study requirements in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-10; Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Response Rate | up to 6 months (180 days)
  95% confidence interval (CI) will be calculated for subjects who achieve Complete response (CR), Partial response (PR), for all AA and MDS subjects, and hematological improvement (HI) for MDS subjects only. Measurement in percentages (%)

SECONDARY OUTCOMES:
Toxicity | study treatment duration (180 days) plus 30 days following last dose of last treatment
  Safety and tolerability parameter monitored according to CTCAE version 4.03 criteria for adverse events and clinical laboratory parameters. Adverse events will be summarized by MedDRA dictionary and by patient population (AA /MDS)
general safety | up to end of study treatment (180 days)
  measurement of vital signs, ECG, and physical exam
tolerability | up to end of end of study treatment (180 days)
  number of subjects who discontinued study treatment early for any reason or due to toxicity
Time to response | up to 5 years
  Interval between treatment start and date of best response following treatment with the BL-8040 in addition to hATG, cyclosporine, and methylprednisolone.
Response duration | up to 5 years
  Time interval between the date of complete response (CR) and the date of first sign of disease recurrence or last follow-up or to the date of last follow-up if patients are alive without disease recurrence, within those patients who have achieved CR.
Overall survival | up to 5 years
  Time from treatment start until the death or last follow-up time (visit or call).
Change in blood product requirements compared to Baseline | up to 6 months (180 days)
  number of transfusions per month compared to Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Tapan Kadia, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States